CLINICAL TRIAL: NCT03811613
Title: Photobiomodulation in Parkinson´s Disease: A Randomized Controlled Trial.
Brief Title: Photobiomodulation and Parkinson
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Luis Santos, Principal Investigator, University of Oviedo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #08/18
Record Dates: First submitted 2019-01-15; First posted 2019-01-22 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2019-01

CONDITIONS: Parkinson Disease
Keywords: movement disorders; light therapy; motor aspects
MeSH Terms: conditions — Parkinson Disease; Movement Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Photobiomodulation group (Experimental): 17 Parkinson´s disease patients were randomly assigned to the photobiomodulation group (experimental group).
  Intervention: Photobiomodulation was administered using red light-emitting diodes (LEDs) with a 670-nm wavelength in six 1-minute blocks alternating the LEDs between the right and left temples, with a 30-second rest between blocks.
  Interventions: Other: Transcranial photobiomodulation
- Sham group (Sham Comparator): 18 Parkinson´s disease patients were randomly assigned to the sham group.
  Intervention: Procedures for the sham group were identical as the photobiomodulation one, except that patients received photobiomodulation during only 5 seconds followed by 55 seconds with no treatment (equalling 1/12th of the energy used for the intervention group).
  Interventions: Other: Transcranial photobiomodulation

INTERVENTIONS:
Other: Transcranial photobiomodulation — Photobiomodulation was administered using red light-emitting diodes (LEDs) with a 670-nm wavelength (which has proven to penetrate the skull)
  Other Names: LEDs

SUMMARY:
This study aimed to assess the effects of transcranial photobiomodulation in patients with Parkinson's disease (PD).

DETAILED DESCRIPTION:
Thirty-five patients with idiopathic PD were randomly assigned to a photobiomodulation (n=17, [mean±SD] 72±7 years) or sham group (n=18, 70±8 years) during 9 weeks (2 sessions/week). The primary endpoint was the motor portion of the Movement Disorders Society-United PD Rating Scale. Secondary endpoints were the Scales for Outcomes in PD, static posturography, walking ability (ten-meter walk test [TMWT]) and functional mobility (timed up and go [TUG] test).

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with idiopathic PD.
* Stage 1-2 on the Hoehn and Yahr Scale.
* Having no neurological condition other than PD.
* Being able to stand for 2 minutes and walk 10 meters without assistance.
* Having no severe dyskinesias or "ON-OFF" phases.

Exclusion Criteria:

- Do not follow inclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
The motor portion of the MDS-UPDRS. | 9 weeks
  The motor portion (part III) Movement Disorders Society-Unified PD Rating Scale. It assesses the motor signs of Parkinson´s disease (minimum and maximum score is 0 and 76 points respectively -the higher score, the higher movement disorder and vice versa-).

SECONDARY OUTCOMES:
Motor function | 9 weeks
  The Spanish-validated version of the Short Parkinson's Evaluation Scale (SPES)/Scales for Outcomes in PD (SCOPA). It measures the Parkinson´s disease patients motor function (minimum and maximum score is 0 and 63 points respectively -the higher score, the worse motor function and vice versa-).
Static posturography | 9 weeks
  The centre of pressure (CoP) parameters (these CoP parameters; Length in mm, Area in mm2 and Speed in m/s are combined to report the static posturography).
Walking speed | 9 weeks
  Ten-meter walk test
TUG | 9 weeks
  Timed up and go test

CONTACTS AND LOCATIONS:
Overall Officials: Luis Santos, PhD, Principal Investigator — Department of Physical Education and Sport (University of León, Spain)
Locations (2):
- Spain (2):
  - Department of Physical Education and Sport, University of León, León, Castille and León
  - University School of Sports Medicine, University of Oviedo, Spain., Oviedo, Principality of Asturias

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Santos L, Olmo-Aguado SD, Valenzuela PL, Winge K, Iglesias-Soler E, Arguelles-Luis J, Alvarez-Valle S, Parcero-Iglesias GJ, Fernandez-Martinez A, Lucia A. Photobiomodulation in Parkinson's disease: A randomized controlled trial. Brain Stimul. 2019 May-Jun;12(3):810-812. doi: 10.1016/j.brs.2019.02.009. Epub 2019 Feb 20. No abstract available. PMID 30824206